CLINICAL TRIAL: NCT05129228
Title: Intraoperative Optical Coherence Tomography of the Saphenous Vein Conduit in Patients Undergoing Coronary Artery Bypass Surgery
Brief Title: Optical Coherence Tomography of the Saphenous Vein Graft
Acronym: OCTOCAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Francis Hospital, New York (Other)
Responsible Party: Principal Investigator, Ziad Ali, MD, DPhil, Director of DeMatteis Cardiovascular Institute, St. Francis Hospital, New York
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-10
Record Dates: First submitted 2021-11-15; First posted 2021-11-22 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Coronary Bypass Graft Stenosis
Keywords: Coronary Artery Bypass Surgery; Saphenous Vein Graft; Intravascular Optical Coherence Tomography; Vein Graft Failure; Coronary Computed Tomography Angiography; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: OCT-guided saphenous vein CABG
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For follow-up visits, in person and via phone, the provider will be blinded. Physicians analyzing Coronary CT Angiograms (CCTA) will be blinded to the randomization arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- OCT-guided saphenous vein graft coronary artery bypass graft surgery (Experimental): Optical Coherence Tomography (OCT) provides high quality intravascular images by using infrared light. OCT will assess the harvested saphenous vein conduit in Coronary Bypass Graft Surgery (CABG). Abnormalities found in the harvested conduits via OCT, at the discretion of the surgeon, will not be utilized for CABG.
  Interventions: Device: OCT-guided saphenous vein CABG
- Visual inspection-guided saphenous vein graft coronary artery graft surgery (No Intervention): Harvested saphenous vein conduits will be assessed visually and will undergo a blinded OCT.

INTERVENTIONS:
Device: OCT-guided saphenous vein CABG — OCT examination of harvested saphenous vein conduits will indicate pathology. Under the surgeon's discretion the conduit segments with pathology will not be grafted.
  Other Names: ILUMIEN OPTIS NEXT OCT Imaging System; ILUMIEN OPTIS OCT Imaging System; OPTIS Integrated OCT Imaging System; OPTIS Mobile OCT Imaging System; Dragonfly Duo Catheter; Dragonfly OPTIS Catheter; Dragonfly OpStar Imaging Catheter; Dual Channel AureFlo Systems; Coronary Flowprobes
  Arms: OCT-guided saphenous vein graft coronary artery bypass graft surgery

SUMMARY:
OCTOCAB is a prospective, randomized (1:1), single-center trial. The purpose of this study is to determine whether intravascular optical coherence tomography (OCT) guided saphenous vein grafting in coronary artery bypass surgery will reduce the rate of early vein graft failure (VGF).

DETAILED DESCRIPTION:
Within the first year of coronary artery bypass grafting (CABG) surgery, the saphenous vein grafts have a failure rate of 10 to 25%. Visual inspection of the vein graft conduit is the current standard in determining the quality of the vein segment. However, there may be intraluminal abnormalities that are undetectable via a visual inspection. OCT examination, using the ILUMIEN OPTIS NEXT OCT Imaging system, of endoscopically harvested saphenous vein conduits will indicate such pathology and enable the surgeon to assess the quality of the harvested vein at the intravascular level.

This study is designed to demonstrate the superiority of OCT-guided saphenous vein CABG in improving the rates of early VGF and the overall outcome of CABG.

The study will follow two randomization arms: OCT-guided saphenous vein CABG (interventional arm) vs. visual inspection-guided saphenous vein CABG (standard of care arm). The analysis of subjects will be with respect to their analyzed group.

Following enrollment, participants will be followed for up to 10 years. The primary endpoint is per graft incidence of vein graft failure. The assessment of the vein graft will be conducted via coronary CT angiogram (CCTA) at 12 months. In the case where the participant has unplanned angiogram due to clinical reasons, prior to the 12 months, the condition of the graft will be determined via the angiogram. Unless all target grafts have reached the endpoint prior to the 12 month time point, a CCTA will be required.

To achieve the power level of 85% at the significance level of 0.025, 760 patients is the anticipated sample size. Analysis will be conducted at the graft level with a Linear Mixed model to account for any potential patient effects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must have evidence of myocardial ischemia (e.g., stable angina, silent ischemia (ischemia in the absence of chest pain or other anginal equivalents), unstable angina, or acute myocardial infarction) suitable for elective CABG.
3. Subject must have undergone coronary angiography identifying at least one lesion that is clinically appropriate and suitable for saphenous vein bypass grafting.
4. Subject must provide written Informed Consent prior to any study related procedure.

Exclusion Criteria:

1. STEMI ≤24 hours from the onset of ischemic symptoms
2. Creatinine clearance ≤30 ml/min/1.73 m2 (as calculated by MDRD formula for estimated GFR) and not on dialysis.
3. Hypotension, shock or need for mechanical support or intravenous vasopressors at the time that the patient would be undergoing the index procedure.
4. CHF (Killip class >2 or NYHA class >3)
5. LVEF <30% by the most recent imaging test within 6 months prior to procedure. If no LVEF test result within 6 months is available, it must be assessed by echocardiography, multiple gated acquisition (MUGA), magnetic resonance imaging (MRI), ventriculography (LV gram) or other method.
6. Unstable ventricular arrhythmias
7. Concomitant multi-valve surgery or major aortic root surgery.
8. Planned non-cardiac surgery within 24 months after the index procedure
9. Prior CABG
10. Any planned PCI within any target vessel(s) within 24 months.
11. Subject has known hypersensitivity or contraindication to any of the study drugs (including aspirin, all P2Y12 inhibitors).
12. Subject has received a heart transplant.
13. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.).
14. Subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy), or the chest/mediastinum.
15. Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
16. Subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
17. Subject has a history of bleeding diathesis or coagulopathy.
18. Subject has life expectancy <2 years for any non-cardiac cause.
19. Pregnant or nursing subjects and those who plan pregnancy in the period up to 2 years following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
20. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Conduit exclusion criteria

1. Severe conduit tortuosity of venous conduit (e.g., with varicosities) such that it is unlikely that the OCT catheter can be delivered without vascular damage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-04-04 (Estimated); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
Vein graft failure (VGF) | 12 months
  Per graft incidence of VGF defined as greater than or equal to 70% in the body of the graft on coronary CT angiography (CCTA)

SECONDARY OUTCOMES:
Target graft failure (TGF) | 12 months
  Composite time-to-first event rate of cardiac death, target graft myocardial infarction (TG-MI), or ischemia-driven target graft revascularization (ID-TGR)
Per graft incidence of ischemic vein graft failure | 12 months
  Greater than or equal to 70% stenosis
Per graft incidence anatomic vein graft failure | 12 months
  Greater than or equal to 50% stenosis
Per patient incidence of vein graft patency | 12 months
  Vein graft having less than 50% stenosis
Per patient incidence of ischemic vein graft failure | 12 months
  Greater than or equal to 70% stenosis
Per patient incidence of anatomic vein graft failure | 12 months
  Greater than or equal to 50% stenosis
Mean vein graft diameter stenosis | 12 months
Mean vein graft area stenosis | 12 months
All-cause mortality | 12 months
Cardiac and non-cardiac mortality | 12 months
All Myocardial Infarction (MI) | 12 months
Target graft myocardial infarction (TG-MI) and Non-Target graft myocardial infarction (non-TG-MI) | 12 months
All revascularization | 12 months
Ischemia driven (ID)-revascularization and Non-ischemia driven (ID)-revascularization | 12 months
Ischemia driven-target graft failure (ID-TGR) | 12 months
Ischemia driven (ID)-revascularization of target native coronary artery subtended by the graft | 12 months

OTHER OUTCOMES:
Intimal injury | 12 months
  Major - Disruption of intima with arc ≥ 60˚ AND length: ≥ 2 mm Minor - Disruption of intima with arc <60˚ AND length: <2 mm
Intraluminal mass | 12 months
  Major - Mass extending ≥ 5 cm and ≥ 2 mm in diameter Minor - Mass extending < 5 cm and < 2 mm in diameter
Intramural hematoma | 12 months
  Major - ≥ 60˚ arc and length ≥ 5mm Minor - < 60˚ arc and length < 5mm
Valvular sclerosis | 12 months
  Major - > 0.25mm thickness Minor - ≤ 0.25mm thickness with redundant valve tissue
Immunohistochemistry | 12 months
  Relationship between the OCT-identified abnormalities with immunohistochemistry in the surplus and OCT-guided excluded segments of vein grafts for histological validation of OCT-identified abnormal findings.
Transit-Time Flow Meter (TTFM) | 12 months
  All grafts will be assessed with TTFM to assess anastomosis. Data will be reviewed to determine whether TTFM abnormalities correlated to OCT findings.
Relationship between OCT parameters and endpoint rates | 12 months
Relationship between OCT parameters at baseline in the standard of care arm with OCT findings in vivo during follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ziad A. Ali, MD,DPhil, Principal Investigator — Saint Francis Hospital; Edward F. Lundy, MD, PhD, Principal Investigator — Saint Francis Hospital
Locations (1):
- St Francis Hospital, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonopoulos AS, Odutayo A, Oikonomou EK, Trivella M, Petrou M, Collins GS, Antoniades C; SAFINOUS-CABG (Saphenous Vein Graft Failure-An Outcomes Study in Coronary Artery Bypass Grafting) group. Development of a risk score for early saphenous vein graft failure: An individual patient data meta-analysis. J Thorac Cardiovasc Surg. 2020 Jul;160(1):116-127.e4. doi: 10.1016/j.jtcvs.2019.07.086. Epub 2019 Aug 26. PMID 31606176
- [Background] Gaudino M, Di Franco A, Bhatt DL, Alexander JH, Abbate A, Azzalini L, Sandner S, Sharma G, Rao SV, Crea F, Fremes SE, Bangalore S. The association between coronary graft patency and clinical status in patients with coronary artery disease. Eur Heart J. 2021 Apr 7;42(14):1433-1441. doi: 10.1093/eurheartj/ehab096. PMID 33709098
- [Background] Caliskan E, de Souza DR, Boning A, Liakopoulos OJ, Choi YH, Pepper J, Gibson CM, Perrault LP, Wolf RK, Kim KB, Emmert MY. Saphenous vein grafts in contemporary coronary artery bypass graft surgery. Nat Rev Cardiol. 2020 Mar;17(3):155-169. doi: 10.1038/s41569-019-0249-3. Epub 2019 Aug 27. PMID 31455868
- [Background] Tan ES, van der Meer J, Jan de Kam P, Dunselman PH, Mulder BJ, Ascoop CA, Pfisterer M, Lie KI. Worse clinical outcome but similar graft patency in women versus men one year after coronary artery bypass graft surgery owing to an excess of exposed risk factors in women. CABADAS. Research Group of the Interuniversity Cardiology Institute of The Netherlands. Coronary Artery Bypass graft occlusion by Aspirin, Dipyridamole and Acenocoumarol/phenoprocoumon Study. J Am Coll Cardiol. 1999 Nov 15;34(6):1760-8. doi: 10.1016/s0735-1097(99)00404-0. PMID 10577567
- [Background] Fitzgibbon GM, Kafka HP, Leach AJ, Keon WJ, Hooper GD, Burton JR. Coronary bypass graft fate and patient outcome: angiographic follow-up of 5,065 grafts related to survival and reoperation in 1,388 patients during 25 years. J Am Coll Cardiol. 1996 Sep;28(3):616-26. doi: 10.1016/0735-1097(96)00206-9. PMID 8772748
- [Background] Goldman S, Copeland J, Moritz T, Henderson W, Zadina K, Ovitt T, Doherty J, Read R, Chesler E, Sako Y, et al. Saphenous vein graft patency 1 year after coronary artery bypass surgery and effects of antiplatelet therapy. Results of a Veterans Administration Cooperative Study. Circulation. 1989 Nov;80(5):1190-7. doi: 10.1161/01.cir.80.5.1190. PMID 2680158
- [Background] Mehta RH, Ferguson TB, Lopes RD, Hafley GE, Mack MJ, Kouchoukos NT, Gibson CM, Harrington RA, Califf RM, Peterson ED, Alexander JH; Project of Ex-vivo Vein Graft Engineering via Transfection (PREVENT) IV Investigators. Saphenous vein grafts with multiple versus single distal targets in patients undergoing coronary artery bypass surgery: one-year graft failure and five-year outcomes from the Project of Ex-Vivo Vein Graft Engineering via Transfection (PREVENT) IV trial. Circulation. 2011 Jul 19;124(3):280-8. doi: 10.1161/CIRCULATIONAHA.110.991299. Epub 2011 Jun 27. PMID 21709060
- [Background] Hattler B, Messenger JC, Shroyer AL, Collins JF, Haugen SJ, Garcia JA, Baltz JH, Cleveland JC Jr, Novitzky D, Grover FL; Veterans Affairs Randomized On/Off Bypass (ROOBY) Study Group. Off-Pump coronary artery bypass surgery is associated with worse arterial and saphenous vein graft patency and less effective revascularization: Results from the Veterans Affairs Randomized On/Off Bypass (ROOBY) trial. Circulation. 2012 Jun 12;125(23):2827-35. doi: 10.1161/CIRCULATIONAHA.111.069260. Epub 2012 May 16. PMID 22592900
- [Background] Raza S, Blackstone EH, Houghtaling PL, Rajeswaran J, Riaz H, Bakaeen FG, Lincoff AM, Sabik JF 3rd. Influence of Diabetes on Long-Term Coronary Artery Bypass Graft Patency. J Am Coll Cardiol. 2017 Aug 1;70(5):515-524. doi: 10.1016/j.jacc.2017.05.061. PMID 28750693
- [Background] Sabik JF 3rd, Lytle BW, Blackstone EH, Houghtaling PL, Cosgrove DM. Comparison of saphenous vein and internal thoracic artery graft patency by coronary system. Ann Thorac Surg. 2005 Feb;79(2):544-51; discussion 544-51. doi: 10.1016/j.athoracsur.2004.07.047. PMID 15680832